CLINICAL TRIAL: NCT06984367
Title: A Socio-Technological Intervention in Community-Based Healthcare for Individuals With Mild Cognitive Impairment (DHEAL-COM-MCI)
Acronym: DHEAL-COM-MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: INRCA_005_2025
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment; Older People
Keywords: social assistive robotics; technology acceptance
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive stimulation arm (Experimental): Daily cognitive stimulation at home with specific software (Brainer) and 1 group session per week, for a total of 12 weeks. Furthermore, each participant will receive the NAO robot at home for a month.
  Interventions: Other: socio-technical intervention
- Control Group (Sham Comparator): Participants in the Control Group will receive a booklet containing information and activities on well-being.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: socio-technical intervention — A daily cognitive stimulation at home with specific software (Brainer) and 1 group session per week. Furthermore, each participant will receive the NAO robot at home.
  Arms: cognitive stimulation arm
Other: Usual care — The subjects will receive a booklet containing information and activities on well-being. They will be invited to do whatever they wish with the information booklet and the proposed exercises, as they would do outside the framework of the experiment. In any case, they will be free to read and do the proposed exercises.
  Arms: Control Group

SUMMARY:
The objectives of the intervention are to counteract the progression of cognitive decline, enhance the intrinsic abilities of users and support the well-being of elderly people with mild cognitive impairment (MCI) through a socio-technical intervention that includes cognitive stimulation, technology and robotics.

DETAILED DESCRIPTION:
The DHEAL-COM-MCI trial is a feasibility pilot with single-blind Randomized Controlled Trial type experimental design. Fifty older adults with Mild Cognitive Impairment (MCI) will be recruited for the study and randomized into two groups: the experimental group, that will perform a stimulation using a specific software, and the control group. Patients in the control group will be offered activities to perform at home, with the same frequency, in line with the usual care activities already proposed by the Neurology Unit. In order to follow the cognitive training, the participants of the Experimental group will receive the following technological devices:

* the software BRAINER, a web platform dedicated to cognitive rehabilitation exercises over 5 different domains such as complex attention, executive function, learning and memory, language and perceptual- motor skills. A dedicated tablet will be provided to the participants to use the Brainer;
* the social robot NAOv6, a fully programmable robot that can interact through its sensors and speech capabilities (i.e RGB camera, ultrasonic proximity sensors on the chest, two microphones, and tactile sensors on the head, hands, feet, and shoulders). NAO is also able to move thanks to multiple joints and actuators, and perform multiple and very complex movements. It can also understand people's language and emotions, as well as respond correctly to any request by speaking and making appropriate gestures;
* In addition, as both NAO and the BRAINER need an internet connection, a webpocket equipped with a SIM card will be given to the user, to allow the 4G connection of the devices. In this way, the functioning of the equipment is guaranteed for the whole period of testing independently of the user's private home/mobile Wi-Fi.

Participants in the Control Group (CG) will receive a booklet containing information and activities on well-being (Appendix A). They will be invited to do whatever they wish with the information booklet and the proposed exercises.

The primary endpoint of the study is to evaluate the perceived stability of the cognitive abilities of older adults with MCI after 12-week of intervention through the MoCA (Montreal Cognitive Assessment) scale.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Mild Cognitive Impairment;
* MoCA ranged 21 - 27;
* Geriatric Depression Scale 5 items (GDS-5items) ≤ 1

Exclusion Criteria:

* Use of active implantable or non-implantable medical devices;
* Nickel allergy;
* Myocardial infarction or stroke within 6 months;
* Painful arthritis, spinal stenosis, amputation, painful foot lesions, or neuropathy that limits balance and mobility;
* Uncontrolled hypertension;
* Pacemaker or implantable cardioverter defibrillator;
* Metastatic cancer or immunosuppressive therapy;
* Significant vision or hearing disturbances.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
cognitive capabilities of older people with MCI | at baseline and 12 weeks later
  It will be assessed through the Montreal Cognitive Assessment (MoCA). The MoCA is a one-page 30-point test administered in approximately 10 minutes. The MoCA assesses several cognitive domains: the short-term memory recall task (5 points), visuospatial abilities (4 points), alternation task (1 point), verbal abstraction task (1 point), attention, concentration, and working memory (6 points), language (6 points), abstract reasoning (2 points), and orientation to time and place (6 points). A score of 26 or above is typically considered within the normal range; scores between 18 and 25 may suggest mild cognitive impairment; scores between 10 and 17 may indicate moderate cognitive impairment; scores below 10 may indicate severe cognitive impairment.

SECONDARY OUTCOMES:
Fragility | at baseline and 12 weeks later
  It will be assessed by the Clinical Frailty Scale (CFS). This descriptive scale divides the older participants into 9 classes based on the information provided by them and their relatives: between 1 and 3 the patient is non-frail, pre-frail if 4, he is frail from 5 to 9.
Health related quality of life | at baseline and 12 weeks later
  The health related quality of life will be evaluated by EQ-5D-5L. The scale consists of five dimensions: mobility, independence, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, mild problems, moderate problems, severe problems and extreme problems. The participant is asked to indicate his/her health status by ticking the box corresponding to the most appropriate statement in each of the five dimensions. The numbers from the five dimensions can be combined into a 5-digit number that describes the health status of the participant. A person reporting "no problems" in all five dimensions would have a health state profile of 11111 (representing full health).
  A person with "slight problems with mobility (2), no problems with self-care (1), moderate problems with usual activities (3), severe pain/discomfort (4), and no anxiety/depression (1)" would have a health state profile of 21341.
  The "worst possible health state" would be 55555.
Psychological Wellbeing | at baseline and 12 weeks later
  The Psychological Wellbeing Scale (PWB) consists of several subscales (self acceptance, positive relationships with others, autonomy, environmental mastery, purpose in life, and personal growth) that measures six aspects of wellbeing and happiness. Individuals respond to the 42 items. Each of the 42 items is rated on a 7-point Likert scale, ranging from 1 ("Strongly disagree") to 7 ("Strongly agree"). The total score can range from 42 to 294, with higher scores indicating greater overall psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Bevilacqua, PhD, Study Chair — IRCCS INRCA, Ancona, Italy
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No